CLINICAL TRIAL: NCT06742034
Title: Translation and Validation of the Visual Analysis of Swallowing Efficiency and Safety Into European Portuguese
Acronym: VASES
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar de Entre o Douro e Vouga (Other)
Collaborators: Aveiro University (Other)
Responsible Party: Principal Investigator, Daniela Ferreira, Speech and Language Pathologist, Centro Hospitalar de Entre o Douro e Vouga
Other Study IDs: 242023
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Deglutition Disorders; Deglutition
Keywords: Dysphagia; Instrumental Assessment; Swallowing Disorders; Fiberoptic Endoscopic Evaluation of Swallow
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to translate and validate to European Portuguese "Visual Analysis of Swallowing Efficiency and Safety - VASES".

ELIGIBILITY:
Inclusion Criteria:

* Patient's FEES recording that allowed good visualization of the pharynx and larynx;
* FEES recording from patients after head and neck surgery who had structural alterations but still did not interfere with a clear visualization of the residues.
* Patient's tracheostomized or under enteral nutrition.

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent FEES at the ULSEDV and met the study's inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Reliable and validated European Portuguese version of the VASES | patients with neurological and/or mechanical oropharyngeal dysphagia evaluated FEES up to 3 months after the first symptomatology
  Visual Analysis of Swallowing Efficiency and Safety (VASES) is a standardized approach for rating pharyngeal residue, penetration, and aspiration during FEES. It establishes clearly defined anatomic and temporal boundaries within which to rate functional swallowing outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Filipa Brás Ferreira, Master, Principal Investigator — Unidade Local de Saúde de Entre Douro e Vouga
Locations (1):
- Centro Hospitalar de Entre Douro e Vouga, Santa Maria da Feira, Portugal